CLINICAL TRIAL: NCT06092580
Title: A Phase 1/2, First-in-human, Open-label Study of Single-agent AWT020 in Patients With Progressive Locally Advanced or Metastatic Cancer
Brief Title: Phase 1 Study of AWT020 in Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anwita Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AWT020-001
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer
Keywords: AWT020; anti-PD1; Interleukine-2; Phase 1; First in human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AWT020 (Experimental): Participants receiving intravenous infusion of AWT020
  Interventions: Biological: AWT020

INTERVENTIONS:
Biological: AWT020 — Participants receiving AWT020 once every two weeks or longer at designated dose levels

SUMMARY:
The aims of this clinical trial are (1) to assess the safety of AWT020 at different dose levels; (2) to determine the pharmacokinetics and pharmacodynamics of AWT020 in subjects with locally advanced or metastatic cancer who have failed standard therapy.

DETAILED DESCRIPTION:
This study will enroll subjects with locally advanced or metastatic cancer who have failed standard therapy. Subjects enrolled into this study will be assigned a dose level and receive AWT020 via intravenous infusion at a regular interval. The treatment will be continued until disease progression, withdrawal from study or death. The primary objective is to investigate the safety of this agent. The secondary objective is to investigate the pharmacokinetics, pharmacodynamic, potential anti-tumor activity and immunogenicity of this agent.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities or procedures.
* Subject must be ≥ 18 years of age or per local regulation.
* Subjects must have a histological diagnosis of solid tumors (carcinoma or sarcoma) or malignant lymphoma, either progressive locally advanced not amenable to local therapy or metastatic, which is refractory, ineligible (in the opinion of the Investigator) or intolerant to standard therapy. Subjects with hepatocellular carcinoma must be diagnosed with dynamic CT or MRI if no tissue diagnosis is available.
* Subject must have performance status of 0, or 1 on the ECOG performance scale.
* Subject with adequate organ function.
* Life expectancy is longer than three months.
* Subject must be able to receive effective contraceptive measures.

Exclusion Criteria:

* Subject is allergic or intolerant to either anti-PD1 or interleukin-2 therapy.
* Subject has received prior immune-check point inhibitors and was discontinued due to greater than grade 3 toxicities.
* Subject is receiving other investigational agent or device.
* Subject has active infection, uncontrolled hypertension, unstable angina, uncontrolled diabetes mellitus, recent myocardial infarction, and congestive heart failure with ejection fraction less than 50%.
* Subject has prior allogeneic stem cell or bone marrow transplant or organ transplant.
* Subject has active central nervous system (CNS) metastases or carcinomatous meningitis.
* Subject with HIV whose viral load is > 400 copies/mL or CD4+ T cell counts are < 350 cells/µL.
* Subject has baseline corrected QT interval (QTc) longer than 480 ms by Fridericia formula.
* Subject is pregnant or breast-feeding.
* Subject has received live virus vaccine within 28 days prior to the first dose of study.
* Any other conditions that might compromise the safety of the subject or the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE 5.0 | From the first infusion up to 90 days after last infusion
  The overall safety of AWT020 in treated subjects

SECONDARY OUTCOMES:
Cmax of AWT020 | 30 minutes after the first infusion in cycle 1 and cycle 2
  The highest serum concentration of AWT020 after infusion
Area under the serum concentration versus time curve (AUC) of AWT020 | First infusion to the end of week 2
  The overall exposure of AWT020 after infusion
Half-life of AWT020 | First infusion to the end of week 2
  The time for the serum concentration of AWT020 to reduce by half
Immunogenicity of AWT020 | Baseline to Cycle 7 Day 1 (each cycle is 28 days)
  The percentage of treated subjects to develop anti-drug antibody against AWT020
Overall response rate in the overall population | During treatment period, an average of 6 months
  The proportion of subjects who achieve a confirmed complete response (CR) or partial response (PR) assessed by investigators
Disease control rate in the overall population | During treatment period, an average of 6 months
  The proportion of treated subjects who have achieved complete response, partial response and stable disease
Progression-free survival in the overall population | 2 years
  The time from the entry of the study until progression or death from any cause, whichever occurs first.
Overall survival in the overall population | 5 years
  The time from the entry of the study to the date of death due to any cause or the date of last contact

CONTACTS AND LOCATIONS:
Overall Officials: Jermaine Coward, BSc (Hons) MBBS MRCP FRACP PhD, Principal Investigator — Icon Cancer Centre South Brisbane
Locations (4):
- Australia (4):
  - ICON Cancer Center South Brisbane, South Brisbane, Queensland
  - Southern Oncology Clinical Research Unit (SOCRU), Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No